CLINICAL TRIAL: NCT00963716
Title: Hot and Cold Biopsy Forceps in the Diagnosis of Endobronchial Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Ajmal khan, Postgraduate Institute of Medical Education and Research
Organization: PIMERIndia (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Khan-1
Record Dates: First submitted 2009-08-18; First posted 2009-08-21 (Estimated); Last update posted 2009-08-21 (Estimated); Status verified 2009-08

CONDITIONS: Endobronchial Growth; Lung Cancer
Keywords: endobronchial biopsy; bronchoscopy; interventional pulmonology
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hot biopsy (Experimental): Hot biopsy i.e. Endobronchial biopsies taken with the application of an electrocoagulation current by an electrocoagulation-capable biopsy forceps
  Interventions: Device: Hot biopsy forceps
- Cold biopsy (Active Comparator): Cold biopsy i.e. Endobronchial biopsies taken without the application of an electrocoagulation current by an electrocoagulation-capable biopsy forceps
  Interventions: Device: Cold biopsy forceps

INTERVENTIONS:
Device: Hot biopsy forceps — Endobronchial biopsies taken with the application of an electrocoagulation current by an electrocoagulation-capable biopsy forceps
  Other Names: Hot biopsy
  Arms: Hot biopsy
Device: Cold biopsy forceps — Endobronchial biopsies taken without the application of an electrocoagulation current by an electrocoagulation-capable biopsy forceps
  Other Names: Cold biopsy
  Arms: Cold biopsy

SUMMARY:
A new electrocautery bronchoscopy biopsy forceps is now commercially available and may prevent bleeding following biopsy. Only one study used this device wherein the authors concluded that the use of hot biopsy forceps for endobronchial biopsy does not appear to have a negative impact on the pathological samples, and that there was a statistically significant, albeit clinically insignificant reduction in bleeding score with hot biopsy forceps. Therefore, a randomized controlled study is required in which the hot and cold biopsies are performed to evaluate the tissue effect of the hot biopsy forceps on histopathological diagnosis.

DETAILED DESCRIPTION:
In recent years, a number of innovative non-thoracotomy techniques have been introduced for the diagnosis of indeterminate pulmonary disease but none has had greater impact on pulmonary medicine than flexible fiberoptic bronchoscopy. Since its introduction in 1968, fiberoptic bronchoscopy has become the procedure of choice for diagnosis and management of many bronchopulmonary disorders. It is accompanied by a low incidence of complications and can be performed satisfactorily by the transnasal approach without general anesthesia. Donlan et al, in 1978, and Ackart and colleagues, in 1983, demonstrated the safety of fiberoptic bronchoscopy as an outpatient procedure.

Transbronchial biopsy was first attempted, through a rigid bronchoscope in 1965, but was associated with a high occurrence of pneumothorax. Reports began to appear from 1974 onwards of lung biopsies done for diffuse pulmonary disease using the standard fiberoptic bronchoscope. Forceps biopsy through flexible bronchoscopy is commonly used to make the cytological or histological diagnosis. Of the procedures performed through bronchoscopy, forceps biopsy provides the best diagnostic yield of 71% to 93%.

A new electrocautery ''hot'' bronchoscopy biopsy forceps is now commercially available and may prevent bleeding following biopsy. Only one study used this device wherein the authors concluded that the use of hot biopsy forceps for endobronchial biopsy does not appear to have a negative impact on the pathological samples, and that there was a statistically significant (albeit clinically insignificant) reduction in bleeding score with hot biopsy forceps. However, limitations in this study were small sample size, use of hot and cold biopsy in the same patient as well as interval between the two biopsies were short due to which it is difficult to decide which technique has contributed to the bleeding. Therefore, a randomized controlled study is required in which the hot and cold biopsies are performed to evaluate the tissue effect of the hot biopsy forceps on histopathological diagnosis.

ELIGIBILITY:
Inclusion Criteria:

1. All patients undergoing routine bronchoscopic biopsy for various indications
2. More than 18 years of age

Exclusion Criteria:

1. Bleeding diathesis
2. On pacemaker or implanted defibrillator
3. On anticoagulation therapy
4. Poor cardiopulmonary reserve
5. Marked hypoxemia
6. Uncooperative patient
7. Enrollment in the previous study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2007-11; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Quality of pathological specimen | 4 hours

SECONDARY OUTCOMES:
Severity of bleeding | During procedure

CONTACTS AND LOCATIONS:
Overall Officials: Ashutosh N Aggarwal, MD, DM, FCCP, Study Chair — PGIMER, Chandigrh
Locations (1):
- Department of Pulmonary Medicine, PGIMER, India, Chandigarh, Uttarakhand, India